CLINICAL TRIAL: NCT07298005
Title: SON4PEM Study: Sonlicromanol in Post-COVID: A Randomized, Double-blind, Placebo-controlled, Phase II Trial
Brief Title: Sonlicromanol in Post-COVID
Acronym: SON4PEM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Michele van Vugt (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Khondrion BV (Industry)
Responsible Party: Sponsor-Investigator, Michele van Vugt, Prof. Dr. M. van Vugt, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-521866-92-01
Record Dates: First submitted 2025-12-11; First posted 2025-12-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Post COVID Condition
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Drug: Sonlicromanol
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sonlicromanol — Sonlicromanol 90mg twice daily for 13 weeks
  Arms: Intervention group
Drug: Placebo — Placebo bid for 13 weeks
  Arms: Placebo group

SUMMARY:
The aim of this randomized, double-blind, placebo-controlled, phase II trial, is to study the effect of sonlicromanol on fatigue in patients with post-COVID who experience post-exertional malaise (PEM).

ELIGIBILITY:
Inclusion Criteria:

* Post COVID according to WHO criteria and verified by post COVID physician
* Post-exertional malaise (PEM) according to DSQ-PEM questionnaire
* Bell's disability score 20-70%
* Mild initial SARS-CoV-2 infection (no hospitalisation)
* WHO performance score of 0 before initial SARS-CoV-2 infection

Exclusion Criteria:

* Patients at risk for cardiac conduction disorders
* History of clinical significant gastro-intestinal surgery or dysmotility that impairs the adsorption of the IMP
* Clinically significant respiratory or cardiovascular disease
* Unstable neurological disease
* Clinically significant active psychiatric disorder that requires treatment
* History of substance abuse
* Active malignancy within the past 5 years
* History of solid organ transplantation
* Active HIV, hepatitis B or C infection
* BMI < 18.5 or > 35
* Pregnancy or breastfeeding
* Clinically relevant laboratory test value outside the reference range
* Use of the following medication, unless stable for at least one month before study and remaining stable throughout the study: (multi)vitamins, co-enzyme Q10, Vitamin E, riboflavin, amino acids, antioxidant supplements and any medication negatively influencing mitochondrial functioning (including but not limited to valproic acid, glitazones, statins, antivirals, amiodarone and NSAIDs)
* Use of the following medication: any moderate or strong Cytochrome P450 (CYP)3A4 inhibitors (all 'conazoles-anti-fungals', HIV antivirals, grapefruit), strong CYP3A4 inducers ((including HIV antivirals, carbamazepine, phenobarbital, phenytoin, rifampicin, St. John's wort, pioglitazone, troglitazone) or any medication metabolized by CYP3A4 with a narrow therapeutic index, medication known to be substrate of Organic Cation Transporter 1 (OCT1) and organic cation transporter 2 (OCT2) or strong P-glycoprotein inhibitors (including amiodarone, azithromycin, captopril, clarithromycin, cyclosporine, piperine, quercetin, quinidine, quinine, reserpine, ritonavir, tariquidar, and verapamil).
* Use of any medication known to affect cardiac repolarization unless QTc interval at screening is normal during stable treatment for a period of two weeks, or 5 half-lives

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Fatigue | Between group differences at week 13
  Post-COVID related fatigue measured with the Fatigue Assessment Scale (FAS), a 10-item questionnaire measuring physical/mental fatigue (ranging from 10-50), with scores <22 indicating no fatigue, 22-34 mild-to-moderate, and ≥35 severe fatigue

SECONDARY OUTCOMES:
Muscle strength | Between group differences at week 13
  Muscle strength measured with the Repeated Handgrip Strength of the dominant hand
Cognitive function | Between group differences at week 13
  Post-COVID related cognitive function measured with the PROMIS cognitive function SF 8a, measures self-perceived cognitive abilities, with scores converted to a T-score (mean 50, SD 10), where higher scores indicate better functioning
Health related quality of life | Between group differences at week 13
  Health related quality of life measured with the SF-36 questionnaire with scores ranging from 0-100, where higher scores indicate better quality of life
Fatigue | Between group differences at week 13
  Post-COVID related fatigue measured with the NeuroQoL SF Fatigue, resulting in a T-score (mean 50, SD 10) where higher scores mean more fatigue

IPD SHARING:
Plan to Share IPD: No